CLINICAL TRIAL: NCT05580016
Title: Prognostic Value of Soluble Urokinase Plasminogen Activation Receptor (SUPAR) to Rule Out Complications in Patients Admitted in Emergency Department for Acute Abdominal Pain.
Acronym: GRADIENT
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GRADIENT
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Soluble Urokinase Plasminogen Activation Receptor; Abdominal Pain; Emergency Department; Mortality
MeSH Terms: conditions — Abdominal Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Soluble Urokinase Plasminogen Activation Receptor measurement
  Interventions: Diagnostic Test: Soluble Urokinase Plasminogen Activation Receptor measurement

INTERVENTIONS:
Diagnostic Test: Soluble Urokinase Plasminogen Activation Receptor measurement — In addition to the standard of care, Soluble Urokinase Plasminogen Activation Receptor levels will be measured in patients.

SUMMARY:
Soluble Urokinase Plasminogen Activation Receptor (SUPAR) is a validated biomarker with applications in the study of inflammation and infection.

Elevated levels of SUPAR have recently been linked to a higher mortality in patients suffering from undifferentiated sepsis, pneumonia, and more recently, COVID-19 infection.

Large randomized controlled trials have been conducted on patients admitted to the emergency department (ER), regardless of the reason for admittance.

These studies have stratified risk based on three cutoffs at initial measurement:

* Low risk : < 3 ng/mL
* Intermediate risk : entre 3 et 6 ng/mL
* High risk : > 6 ng/mL Low levels of SUPAR are associated with low risk of mortality in the short and long term in patients presenting to the ED, no matter the reason for admittance. Risk stratification could be an added decision-making tool for clinicians to comfort hospital discharge.

To the best of our knowledge, there is no available data on the added value of SUPAR for predicting mortality in abdominal sepsis and abdominal pain.

Abdominal pain is responsible for 10 to 30 % of ER admissions. Consequently, abdominal pain is then responsible for roughly 10 % of admissions into medical and surgical wards. Mortality varies depending on patient factors. Mortality is usually stratified on age. In patients under 50 years of age, it is near 8%, but it reaches 19 % in patients over 50.

Diagnostic accuracy also decreases drastically with age, reaching approximately 30 % patients over 75.

Taking this into account, integrating a measure of SUPAR levels into the current standard of care could stratify the risk of complications in patients admitted to the ER with abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Over 18 years of age
* Presenting to the ED with abdominal pain for over an hour
* Classified as category 2 or above on the CIMU or FRENCH severity scale
* Necessitating bloodwork at the discretion of the consulting physician
* Who gave his Non-opposition after clear and fair information on the study

Exclusion Criteria:

Patients :

* With pain evocative of kidney stones
* With a chronic inflammatory disease: HIV infection, inflammatory bowel disease, rheumatoid arthritis, cancer
* Chronic renal disease
* Under hospice care
* Intubated
* Unstable hemodynamically
* Transferred from a secondary care facility and having undergone previous bloodwork
* Patient unable to understand the information and to give his non-objection
* under guardianship, curatorship or subordination;
* benefiting from enhanced protection, namely: minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in an establishment health or social, adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the emergency department for abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of medical and surgical complications within 7 days | 7 days
  7 -day complications as a composite outcome of either:
  * Necessity of surgical intervention
  * Hospitalisation lasting over 24 hours
  * Death in direct relation to the reason for admittance
  * Hospital readmission for abdominal pain in a similar abdominal quadrant

SECONDARY OUTCOMES:
Occurrence of medical and surgical complications within 30 days | 30 days
  30 -day complications as a composite outcome of either:
  * Necessity of surgical intervention
  * Hospitalisation lasting over 24 hours
  * Death in direct relation to the reason for admittance
  * Hospital readmission for abdominal pain in a similar abdominal quadrant
Optimal cutoff | 7 days
  Determining optimal cutoffs for Soluble Urokinase Plasminogen Activation Receptor through Area Under Curve using Receiver Operating Characteristic method for patients presenting complications of abdominal pain in the first seven days.
Comparison with routine biomarkers | 30 days
  Comparison of diagnostic performance with other routine biomarkers:
  Procalcitonine C-Reactive Protein Lactate

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Poitiers, Poitiers, France